CLINICAL TRIAL: NCT05655208
Title: Histological Profiles of Lung Allograft Transbronchial Biopsies and Clinical Outcomes After Lung Transplantation
Acronym: LANDSCAPE
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Collaborators: Hopital Foch (Other)
Responsible Party: Sponsor
Other Study IDs: LungCluster
Record Dates: First submitted 2022-11-29; First posted 2022-12-19 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Lung Transplant Rejection
Keywords: Lung transplantation; Rejection; Transbronchial biopsy; Donor specific Antibody; Cluster analysis
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung transplantation is the only curative treatment for individuals with end-stage lung disease. Understanding the lung allograft's histological lesions, which is key for the patient management, remains difficult because of the multiplicity of lesions associated with graft outcome and their interpenetration.

The goal of this observational study is to identify clusters of histological lesion on transbronchial biopsies in Lung transplant recipient prospective cohort.

The main question[s] it aims to answer are:

* what are the different pattern of histological lesion?
* what are the graft outcome associated with the different clusters?

DETAILED DESCRIPTION:
SCIENTIFIC JUSTIFICATION:

With more than three million deaths per year, the chronic obstructive pulmonary disease is currently the third cause of mortality worldwide , and contributes to the growing number of individuals with end-stage lung disease, which is now a major issue for world public health. Overall, for individuals with end-stage lung disease, lung transplantation (LTx) is the only treatment able to increase patient survival and quality of life, with more than 4,500 lung transplantations performed each year.

Despite major progresses made in the last decade regarding organ preservation, procurement and short term outcome little improvements have been made on the histological characterization of rejection, which remains the main determinant of patient death after lung transplantation.

One of the main limitation of histological analysis is the multiplicity of lesions associated with graft outcome and their interpenetration. Historically, the perivascular infiltrate or cellular rejection (A lesions), and the lymphocytic bronchiolitis (B lesions) are the first histological lesions associated with graft dysfunction and stand as key parameters in patient management. In addition to A and B lesions, a wide spectrum of histological lesions of the lung allograft is associated with clinical outcomes.

However, to our best knowledge, only few studies thoroughly investigated the various elementary lesions in the broad scope of histological analysis, and their association with clinical outcomes. Although informative, those studies usually suffer from a small number of patients, convenience clinical samples from registry, and the lack of innovative statistical approach. Overall, the wide spectrum of the allograft lesions has not been investigated using a large number of transbronchial biopsies with standardized protocol and biopsy reading, and a multidimensional approach on deeply phenotyped data.

The recent use of unsupervised method in organ transplantation has permitted the identification of clinically relevant patient clusters and may be a relevant strategy to decipher the heterogeneity in histological lesions in lung recipients.

Therefore, using a deeply phenotyped prospective cohort of lung recipients and consecutive transbronchial biopsies with protocolized evaluation and interpretation covering the different cases scenario encountered in clinical practice, the investigators aim to identify histological clusters based on histological lesions and assess their associations with graft and patient outcomes.

OBJECTIVES:

Main objective: To identify of histological cluster of lung allograft Transbronchial biopsies

Secondary objective: To evaluate association of each cluster with baseline clinical data and anti HLA donor specific antibody and graft outcome

INTERVENTIONS:

This is an observational study that involves only minimal risk and constraints. The intervention consists in the evaluation of parameters measured as part of the standard of care at the time of post-transplant allograft biopsy.

No medicinal product is under investigation in this protocol.

EXPECTED BENEFITS for the participants and for society:

There will be no immediate individual benefit for the patient to participate in the study.

This study will provide us with data of Lung transplant patients that may allow the improvement of clinical decisions and the long-term lung allograft management.

MINIMAL RISKS AND CONSTRAINTS added by the study No additional intervention beyond the standard of care will be performed in this study.

RECRUITING CENTER:

* Single center study
* Hopital Foch, Suresnes, France

ELIGIBILITY:
Inclusion Criteria:

* i) age greater than 18 years,
* ii) single or bilateral lung transplantation,
* iii) having at least one transbronchial biopsy available for analysis
* iv) consent their clinical data to be used for research

Exclusion Criteria:

• Biopsies with at least one missing value in the standardized clinical report were excluded

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective cohort included consecutive lung transplant recipients who were transplanted between February 2010 and November 2019 in Foch Hospital and were eligible for inclusion.
  Every protocol and for cause transbronchial biopsies (TBBs) identified in the Foch hospital database for each patient were analyzed using standardized template. Reports of TBB with one or more missing values were excluded. Protocol TBB were performed after transplantation with the following scheme : month 1 (M1) at 30 ± 10 days, month 2 (M2): 60 ± 10 days, month 3 (M3): 90 ± 10 days, month 4 (M4): 120 ± 10 days, month 6 (M6): 180 ± 10 days, month 9 (M9): 270 ± 10 days and month 12 (M12): 365 ± 10 days. For cause TBB were performed in case of graft dysfunction.
Sampling Method: Non-Probability Sample
Enrollment: 498 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
graft loss resulting in death or re-transplantation and all-cause mortality | 118 months

SECONDARY OUTCOMES:
chronic lung allograft dysfunction occurrence | 118 months

IPD SHARING:
Plan to Share IPD: Yes
We will agree to share IPD under reasonnable request and for research purpose only. Any request should be send to Pr Roux Antoine at the following email adress: rouxantoine@hotmail.com
Supporting Information: Study Protocol, SAP, ICF